CLINICAL TRIAL: NCT05407831
Title: Lean Diabetes Study
Status: Withdrawn | Type: Observational
Why Stopped: Per Endocrinology study team, COVID prevented enrollment, and then PI left institution.
Sponsor: Leon Fogelfeld MD (Other Government)
Responsible Party: Sponsor-Investigator, Leon Fogelfeld MD, Principal Investigator, Cook County Health
Organization: Cook County Health (Other Government)
Other Study IDs: 19-204
Record Dates: First submitted 2022-06-02; First posted 2022-06-07 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Lean Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Saliva collection
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- LDM: Lean Diabetes Mellitus
  Interventions: Genetic: Genetic; Behavioral: Social habits; Other: Perinatal stress
- ODM: Obese Diabetes Mellitus
  Interventions: Genetic: Genetic; Behavioral: Social habits; Other: Perinatal stress

INTERVENTIONS:
Genetic: Genetic — Calculate MODY probability
Behavioral: Social habits — Alcohol vs Smoking vs Drug use
Other: Perinatal stress — Survey

SUMMARY:
Systematic assessment of perinatal, behavioral and genetic risk factors will be evaluated in an underserved population with lean diabetes (LDM) as compared to a control population with obese type 2 diabetes (ODM).

DETAILED DESCRIPTION:
Background:

The prevalence of lean (BMI <25, non-type 1) diabetes (LDM) is not rare; however, the reason why these individuals develop diabetes without traditional risk factors is often not investigated. Since this subset of individuals with diabetes are not overweight, they represent an ideal population to examine the causes of diabetes development without the confounding effect of obesity. Understanding critical risk factors for non-autoimmune causes of beta cell underdevelopment, injury and failure can impact prevention, early detection and even treatment in this population of lean individuals. Guidelines for diabetes management currently mainly targets either type 1 or overweight/obese type 2 diabetes (ODM) with a lack of guidance on how best to personalize work-up and treatment in LDM.

Objective:

Systematic assessment of perinatal, behavioral and genetic risk factors will be evaluated in an underserved population with LDM as compared to a control population with ODM. Understanding why certain lean individuals develop diabetes will potentially elucidate mechanisms that could be masked when obesity is also present.

Study Hypothesis:

LDM patients have more impaired beta cell function than classic ODM. The potential pathogenic drivers for the beta-cell impairment in LDM may involve in-utero/childhood malnutrition, lifestyle insults to beta-cells like alcohol and smoking and specific genetic traits that impair beta cell function.

ELIGIBILITY:
Inclusion Criteria:

Cases: BMI <25 with diabetes, not having exclusion criteria Controls: BMI >29 with diabetes, not having exclusion criteria

Exclusion Criteria:

individuals <20 years of age, currently pregnant or undergoing chemotherapy, those on glucocorticoid therapy; history of bariatric surgery or pancreatitis; known positive antipancreatic antibodies; individuals with a BMI between 25.0-29.9, A1c >10%

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 35 adults with LDM (BMI <25) will be compared to age, gender and duration of diabetes matched control population of 35 ODM (BMI >30) adults recruited from the CCH outpatient clinics.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2023-07-26 (Actual); Study Completion 2023-07-26 (Actual)

PRIMARY OUTCOMES:
HOMA Index and Beta cell function | Single visit study

SECONDARY OUTCOMES:
Prevalence of high risk behaviors | Single visit study
Prevalence of perinatal malnutrition | Single visit study
MODY probability >25% | Single visit study

CONTACTS AND LOCATIONS:
Locations (1):
- Cook County Health, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No